CLINICAL TRIAL: NCT01277497
Title: A Randomized Study on the Effects of Sevelamer Carbonate Versus Calcium Acetate on Biomarkers of Vascular Calcification, Inflammation, and Endothelial Dysfunction in Chronic Kidney Disease Stages 3 and 4
Brief Title: Effect of Phosphate Binders on Markers of Vascular Health in Chronic Kidney Disease Stages 3 and 4
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Albany College of Pharmacy and Health Sciences (Other)
Collaborators: Albany Medical College (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Darius Mason, PI, Albany College of Pharmacy and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2902
Record Dates: First submitted 2011-01-06; First posted 2011-01-17 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Phosphate binder; Sevelamer carbonate; Calcium acetate; Vascular calcification; Endothelial Dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vascular Calcification | interventions — Sevelamer; calcium acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevelamer carbonate (Experimental): 1,600 mg (2 x 800 mg) three times daily with meals for a total of 12 weeks
  Interventions: Drug: Sevelamer carbonate
- Calcium acetate (Active Comparator): 1,334 mg (2 x 667 mg) three times daily with meals for a total of 12 weeks
  Interventions: Drug: Calcium acetate

INTERVENTIONS:
Drug: Sevelamer carbonate — Sevelamer carbonate 1,600 mg three times daily with meals
  Other Names: Renvela
  Arms: Sevelamer carbonate
Drug: Calcium acetate — Calcium acetate 1,334 mg three times daily with meals for 12 weeks
  Other Names: Phoslo
  Arms: Calcium acetate

SUMMARY:
Chronic kidney disease (CKD) patients often have high levels of a substance called fibroblast growth factor-23 (FGF-23), a phosphorus excreting hormone, which has been related to heart disease. As kidney function declines, less phosphorus is removed by the kidneys and as a result phosphorus accumulates in the blood. In response to elevated phosphorus levels, more FGF-23 is released to help facilitate the excretion of extra phosphorus into the urine. In addition to effects on FGF-23, increased phosphorus levels can lead to calcification (hardening) of the blood vessels in the CKD population.

Phosphate binding medicines are used in CKD patients to lower the amount of phosphorus absorbed by the stomach and intestines after eating meals and snacks. In patients with CKD, studies have shown that phosphate binders can lower FGF-23 levels in the blood. Lowering FGF-23 levels in CKD patients may also lower substances in the blood that cause calcification of blood vessels in the CKD population.

This study is being done to determine if using phosphate binders, either sevelamer carbonate or calcium acetate, in the earlier stages kidney disease (before dialysis) can decrease FGF-23 and biomarkers (substances in the blood) associated with hardening of the blood vessels and heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 18 years of age at start of screening
* CKD stage 3 or 4 defined by an eGFR 15 - 60 mL/min/1.73m2
* Not expected to start dialysis for 8 months
* Serum intact PTH < 500 pg/mL during screening period
* On a stable ACE inhibitor/ARB regimen for 30 days prior to screening

Exclusion Criteria:

* History of any of the following diseases: congestive heart failure, MI within the last 6 months, cerebrovascular accident, significant valvular disease, malignancy
* Currently receiving erythropoiesis stimulating agent or IV iron therapy
* History of inflammatory/autoimmune disease
* History of polycystic kidney disease
* HIV positive or AIDS
* Pregnant or breastfeeding
* Receiving activated Vitamin D analogs, nutritional vitamin D agents > 2,000 IU/day, or calcimimetics with in the last 3 months
* Significant GI disorder
* Proteinuria >3.5 g/24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the change in FGF-23 concentrations | 12 weeks

SECONDARY OUTCOMES:
Change in vascular calcification biomarker levels | 12 weeks
Change in endothelial dysfunction biomarker levels. | 12 Weeks
Change in inflammatory biomarker levels | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Darius L Mason, Pharm.D., Principal Investigator — Albany College of Pharmacy and Health Sciences
Locations (1):
- Albany Medical Center South Clinical Campus, Albany, New York, United States

REFERENCES:
- [Derived] Mason DL, Godugu K, Nnani D, Mousa SA. Effects of sevelamer carbonate versus calcium acetate on vascular calcification, inflammation, and endothelial dysfunction in chronic kidney disease. Clin Transl Sci. 2022 Feb;15(2):353-360. doi: 10.1111/cts.13151. Epub 2021 Oct 2. PMID 34599865